CLINICAL TRIAL: NCT05288517
Title: Firearm Safe Storage Decision Aid for Adults With Suicide Ideation
Brief Title: A Randomized Control Trial of a Digital Health Tool
Acronym: L2L
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1477456
Record Dates: First submitted 2022-03-10; First posted 2022-03-21 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Suicide and Self-harm
MeSH Terms: conditions — Suicide; Self-Injurious Behavior

STUDY DESIGN:
Intervention Model Description: Patients identified as at risk for suicide using a prediction model were randomized using a 1:1 allocation to receive invitation to visit Lock to Live (L2L) or control.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (No Intervention): Control patients received three invitations for a survey only and were blind to the L2L intervention.
- Lock to Live Intervention Arm (Active Comparator): Patients in the Intervention Arm received the invitation to Lock to Live, including up to 3 EHR invitation messages plus three messages to complete a follow-up survey evaluating study outcomes.
  Interventions: Behavioral: Lock to Live

INTERVENTIONS:
Behavioral: Lock to Live — Lock to Live is an anonymous web-based self-administered decision aid for safe firearm and medication storage (Public URL: http://lock2live.com/).
  Arms: Lock to Live Intervention Arm

SUMMARY:
This randomized trial evaluated whether sending population-based invitation messages through the electronic health record to visit Lock to Live (L2L), a web-based decision aid that incorporates patients' values into recommendations for safe storage of firearms and medications, impacted readiness to change firearm and medication storage behaviors.

DETAILED DESCRIPTION:
Lock to Live (L2L) is a web-based decision aid that incorporates patients' values into recommendations for safe storage of firearms and medications. This randomized trial evaluated whether sending population-based invitation messages to visit L2L through the Electronic Health Record (EHR) to patients treated in primary care and mental health specialty settings with elevated suicide risk, identified using a prediction model, impacted readiness to change firearm and medication storage behaviors.

Patients were identified using previously validated suicide risk prediction models developed within the Mental Health Research Network (MHRN). These models are highly predictive of suicide attempt and death by suicide for both a 30-day and 90-day period. Patients in the 75-99.5th risk percentiles were randomized. Half were randomized to receive L2L+survey (intervention) and half received survey only (control).

and control groups. Over 21,000 unique patients were enrolled over a 6-month period.

Survey respondents were assigned to one of five groups based on readiness for change: pre-contemplative (do not believe in safe storage), contemplative (believe in safe storage but not doing it), thinking (considering changing storage), preparation (planning to change storage), or action (safely storing). Data will be analyzed using chi-square, logistic and multinomial logit models to test for differences between intervention and control groups.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or older (>18 yrs.)
* suicide risk based on validated risk algorithm (patients falling within the 75th- 99th risk percentile based on the suicide risk algorithm)
* Patients with a recent visit within Mental Health department or within Primary Care department w. Mental Health diagnosis (recent defined as within the prior month from the date of the algorithm run date)
* English noted as primary language, or patient flag for interpreter needed is not set
* Patient is not deceased
* Patient is registered on kp.org to receive online message

Exclusion Criteria:

* A recorded diagnosis of: Dementia/ or other cognitive impairment (including developmental delay), Psychosis, Schizophrenia, Autism Spectrum Disorder
* Non-English speaker
* Receiving home-based palliative care, or hospice care
* In a skilled nursing facility
* On the Research Exclusion list - Do Not Contact
* Patient has flag for health proxy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20131 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Anonymous Survey measuring Change Readiness developed after Prochaska and DiClemente's stage of change theory. | Between 2 weeks and 4 weeks following invitation to Lock to Live intervention.
  Patient reported readiness to change safe storage behavior for firearms and medications.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer M Boggs, PhD, Principal Investigator — Institute for Health Research, Kaiser Permanente Colorado
Locations (1):
- Kaiser Permanente Colorado, Institute for Health Research, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Betz ME, Kautzman M, Segal DL, Miller I, Camargo CA Jr, Boudreaux ED, Arias SA. Frequency of lethal means assessment among emergency department patients with a positive suicide risk screen. Psychiatry Res. 2018 Feb;260:30-35. doi: 10.1016/j.psychres.2017.11.038. Epub 2017 Nov 14. PMID 29169036
- [Background] Diurba S, Johnson RL, Siry BJ, Knoepke CE, Suresh K, Simpson SA, Azrael D, Ranney ML, Wintemute GJ, Betz ME. Lethal Means Assessment and Counseling in the Emergency Department: Differences by Provider Type and Personal Home Firearms. Suicide Life Threat Behav. 2020 Oct;50(5):1054-1064. doi: 10.1111/sltb.12649. Epub 2020 Jun 29. PMID 32598076
- [Background] Betz ME, Knoepke CE, Siry B, Clement A, Azrael D, Ernestus S, Matlock DD. 'Lock to Live': development of a firearm storage decision aid to enhance lethal means counselling and prevent suicide. Inj Prev. 2019 Sep;25(Suppl 1):i18-i24. doi: 10.1136/injuryprev-2018-042944. Epub 2018 Oct 13. PMID 30317220
- [Background] Simon GE, Rutter CM, Peterson D, Oliver M, Whiteside U, Operskalski B, Ludman EJ. Does response on the PHQ-9 Depression Questionnaire predict subsequent suicide attempt or suicide death? Psychiatr Serv. 2013 Dec 1;64(12):1195-202. doi: 10.1176/appi.ps.201200587. PMID 24036589
- [Derived] Boggs JM, Quintana LM, Beck A, Clarke CL, Richardson L, Conley A, Buckingham ET, Richards JE, Betz ME. A Randomized Control Trial of a Digital Health Tool for Safer Firearm and Medication Storage for Patients with Suicide Risk. Prev Sci. 2024 Feb;25(2):358-368. doi: 10.1007/s11121-024-01641-6. Epub 2024 Jan 11. PMID 38206548
- See also: Decision-aid tool for safer firearm and medication storage — https://lock2live.org/